CLINICAL TRIAL: NCT03255044
Title: Impact of Lipophilic Versus Hydrophilic Statin Administration on The Clinical Outcome and Cardiac Markers of Patients With Heart Failure
Brief Title: Comparison of Lipophilic Versus Hydrophilic Statins on Patients With Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nouran Omar, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 48
Record Dates: First submitted 2017-08-10; First posted 2017-08-21 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: statin; hydrophilic; lipophilic
MeSH Terms: conditions — Heart Failure | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lipophilic statin (Active Comparator): Atorvastatin 40 mg administered daily in addition to guideline directed therapy for heart failure.
  Interventions: Drug: Atorvastatin; Other: guideline directed therapy
- Hydrophilic statin (Active Comparator): Rosuvastatin 20 mg administered daily in addition to guideline directed therapy for heart failure.
  Interventions: Drug: Rosuvastatin; Other: guideline directed therapy

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin administered as well as standard heart failure therapy
  Other Names: standard heart failure therapy
  Arms: Lipophilic statin
Drug: Rosuvastatin — Rosuvastatin administered as well as standard heart failure therapy
  Other Names: standard heart failure therapy
  Arms: Hydrophilic statin
Other: guideline directed therapy — standard heart failure therapy

SUMMARY:
There is a controversy whether statins are beneficial in patients with heart failure or not. Trials in which lipophilic statins have been used revealed positive results, unlike major studies where hydrophilic statins were administered. This trial is designed to compare the effects of lipophilic versus hydrophilic statin use in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years (of both sexes)
* diagnosed with stable chronic heart failure NYHA class II-III
* ejection fraction < 40 % as assessed by 2D echocardiography
* who have been optimized on Guideline Directed treatment for heart failure for at least a month prior to enrolling.

Exclusion Criteria:

* Known hypersensitivity to statin
* Treatment with statins during the past month prior to study.
* Serum creatinine > 3 mg/dl
* Significant liver disease: liver enzymes 2.5 folds the upper normal limit
* Malignancy
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction (LVEF) | 6 months
Left Ventricular End-diastolic volume (LVEDV) | 6 months
Left Ventricular End-systolic volume (LVESV) | 6 months
cardiac markers | 6 months
  NT pro BNP (N-terminal prohormone of brain natriuretic peptide) sST2 (soluble suppression of tumorigenicity 2)

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire( MLHFQ) | 6 months
Packer composite outcome | 6 months
  * Patients are considered improved if at the final visit they experienced a favorable change in NYHA functional class or in the patient global assessment: markedly/moderately improved (or both) but did not experience any major adverse clinical events during the course of the trial (death or hospitalization).
  * Patients are considered worse if they experienced a major clinical event during the duration of treatment or reported worsening of their NYHA class or global assessment at the final visit.
  * Patients are considered unchanged if they are neither improved nor worse.

OTHER OUTCOMES:
Incidence of major adverse cardiac events | 6 months
  * Cardiovascular death
  * All cause death
  * Non- fatal myocardial infarction
  * Stroke
Incidence of Hospitalization | 6 months
  Defined as hospitalization for worsening of heart failure for more than 24 hours and demanding aggressive intervention (IV inotropics, diuretics etc..)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital Cardiology Rehab Unit, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El Said NO, El Wakeel LM, Khorshid H, Darweesh EAG, Ahmed MA. Impact of lipophilic vs hydrophilic statins on the clinical outcome and biomarkers of remodelling in heart failure patients: A prospective comparative randomized study. Br J Clin Pharmacol. 2021 Jul;87(7):2855-2866. doi: 10.1111/bcp.14695. Epub 2021 Jan 3. PMID 33294980